CLINICAL TRIAL: NCT02953041
Title: The Effect of Glycopyrronium and Indacaterol, as Monotherapy and in Combination, on the Methacholine Dose-response Curve
Brief Title: Effect of a LAMA and a uLABA on the Methacholine Dose-response Curve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, MD, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MCh-DRC-1
Record Dates: First submitted 2016-10-24; First posted 2016-11-02 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Glycopyrrolate; indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAMA Treatment (Experimental): Inhalation of 50mcg glycopyrronium from Breezhaler device 1 hour prior to methacholine challenge
  Interventions: Drug: Glycopyrronium
- uLABA Treatment (Experimental): Inhalation of 75mcg indacaterol from Breezhaler device 1 hour prior to methacholine challenge
  Interventions: Drug: Indacaterol
- Combo Treatment (Experimental): Inhalation of 50mcg glycopyrronium from one Breezhaler device, and 75mcg indacaterol from a second Breezhaler device, all one hour prior to methacholine challenge
  Interventions: Drug: Glycopyrronium; Drug: Indacaterol

INTERVENTIONS:
Drug: Glycopyrronium — long-acting muscarinic antagonist
  Other Names: Seebri, Glycopyrrolate, Glycopyrronium bromide
  Arms: Combo Treatment; LAMA Treatment
Drug: Indacaterol — ultra long-acting beta agonist
  Other Names: Onbrez
  Arms: Combo Treatment; uLABA Treatment

SUMMARY:
The study will assess the effects of two drugs, glycopyrronium and indacaterol, taken either as monotherapy or in combination, on the methacholine dose-response curve. This will allow for further elucidation of the mechanisms of each drug in human participants.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, three-way crossover study testing glycopyrronium (Seebri®) vs. indacaterol (Onbrez®) vs. glycopyrronium+indacaterol. The MCT method used will be the two-minute tidal breathing dosing protocol. The investigators plan to enroll thirty participants, fifteen asthmatics and fifteen non-asthmatics participants.

* Asthmatic Participants Procedure: Each participant will undergo a total of twelve MCh challenges. Each MCh challenge will be stopped when the response to MCh reaches a plateau, when the participant's FEV1 drops 40% from baseline, when the highest concentration of MCh (128mg/mL) has been administered, or if the participant wishes to stop (e.g. due to discomfort). For the purpose of this study, a plateau will be defined as the last 3 consecutive data points falling within 5%. The first day of testing will take approx. 3hrs. and will entail participants undergoing a MCh challenge to determine their baseline MCh PC20. They will then self-administer the contents of two Breezhaler inhalers. If taking one of the monotherapies, one inhaler will contain active treatment (50mcg glycopyrronium or 5mcg indacaterol) and the other inhaler will contain a placebo. For the combination treatment arm, both inhalers will contain active drug (one 50mcg glycopyrronium and one 75mcg indacaterol). The identity of the treatment administered will be unknown to the participants and to the study staff. Participants will then undergo MCT post-treatment at 1 hr., 24 hrs., and 48 hrs. Testing at 24 and 48 hrs. will take approximately 1-1.5 hrs. Therefore, participants must attend the lab at roughly the same time of day for three consecutive days for each treatment arm. Following a minimum 10-day washout between treatment administrations, the same procedure will be repeated with the second study treatment. Following a second 10-day washout, the procedure will be repeated with the third study treatment.
* Non-Asthmatic Participants Procedure: Each non-asthmatic participant will undergo a single MCh challenge, which should take approx. 1-1.5 hrs. This will allow for the generation of a "normal" MCh DRC curve to compare with the asthmatic data. The MCh challenge will be stopped when the response to MCh reaches a plateau, when the participant's FEV1 drops 40% from baseline, when the highest concentration of MCh (128mg/mL) has been administered, or if the participant wishes to stop.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 or older
* stable mild-to-moderate asthma
* baseline methacholine PC20 less than or equal to 8mg/mL and FEV1 greater than or equal to 65% of predicted (asthmatic participants)
* baseline methacholine PC20 greater than 16mg/mL (healthy participants)

Exclusion Criteria:

* use of long-acting bronchodilators or long-acting muscarinic antagonists within 30 days of Visit 1
* pregnant or lactating
* cardiovascular, prostate, kidney or urinary retention problems
* respiratory illness within 4 weeks of Visit 1
* allergen-induced asthma exacerbating within 4 weeks of Visit 1
* hypokalemia
* diabetes
* glaucoma
* smokers and exsmokers with greater than 10 pack years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline methacholine bronchoprotection at 1 hour | baseline versus 1 hour post-treatment
  assessed by dose shift of geometric mean methacholine PC20 data

SECONDARY OUTCOMES:
Change from baseline methacholine bronchoprotection at 24 hours | baseline versus 24 hours post-treatment
  assessed by dose shift of geometric mean methacholine PC20 data
Change from baseline methacholine bronchoprotection at 48 hours | baseline versus 48 hours post-treatment
  assessed by dose shift of geometric mean methacholine PC20 data

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
Journal Publication

REFERENCES:
- [Derived] Blais CM, Davis BE, Cockcroft DW. The effect of glycopyrronium and indacaterol, as monotherapy and in combination, on the methacholine dose-response curve of mild asthmatics: a randomized three-way crossover study. Respir Res. 2017 Aug 2;18(1):146. doi: 10.1186/s12931-017-0628-4. PMID 28768531